CLINICAL TRIAL: NCT01412463
Title: DURABILITY+ : a Prospective, Multi-center, Controlled Study Measuring the Durability in Lesions of the Superficial Femoral Artery of the Protégé Everflex+ Stent
Brief Title: DURABILITY+ : a Prospective, Multi-center, Controlled Study With the Everflex+ Stent in SFA Lesions
Acronym: DURABILITY+
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Flanders Medical Research Program (Network)
Collaborators: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMRP-101208
Record Dates: First submitted 2011-08-08; First posted 2011-08-09 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Protégé EverFlex+ (Experimental): Stenting with Protégé EverFlex+
  Interventions: Device: stent placement

INTERVENTIONS:
Device: stent placement — * pre-dilation of the study lesion is mandatory
  * stent placement with 1 Protégé Everflex+ stent
  * only 1 stent is allowed within the study protocol
  * post-dilation may be performed but is not mandatory
  Other Names: Protégé EverFlex+

SUMMARY:
The objective of this study is to evaluate the immediate and long-term (up to 12 months) safety and effectiveness of primary stenting with the Protégé Everflex+ stent system for the treatment of superficial femoral artery (SFA) lesions (without involvement of the popliteal artery) between 40 mm and 180 mm in length.

ELIGIBILITY:
General Inclusion Criteria:

* De novo, restenotic or reoccluded (from PTA or adjunct therapy, not including stents or stent grafts) lesion located in the superficial femoral artery (without popliteal involvement) with proximal point at least one centimeter below the origin of the profunda femoralis and suitable for stenting
* Patient presenting with a score from 2 to 4 following Rutherford classification
* Patient is willing to comply with specified follow-up evaluations at the specified times
* Patient is >18 years old
* Patient (or their legal representative) understands the nature of the procedure and provides written informed consent, prior to enrollment in the study

Angiographic Inclusion Criteria

* The length of the target lesion is minimally 40 mm and maximally 180 mm, to be covered with one stent
* The target lesion has angiographic evidence of stenosis or restenosis > 50% or occlusion which can be passed with standard guidewire manipulation
* Target vessel diameter visually estimated is >3.5 mm and <7.5 mm
* Prior to enrollment, the guidewire has crossed target lesion
* There is angiographic evidence of at least one-vessel-runoff to the foot, irrespective of whether or not outflow was re-established by means of previous endovascular intervention
* Patient is eligible for treatment with the Protégé Everflex+ stent system

General Exclusion Criteria:

* Presence of another stent or stent graft in the target vessel that was placed during a previous procedure
* Previous by-pass surgery in the same limb requiring access to the target lesion
* Patients for whom antiplatelet therapy, anticoagulants or thrombolytic drugs are contraindicated or no alternative is available
* Patients with known hypersensitivity to nickel-titanium
* Patients with uncorrected bleeding disorders
* Female patient with child bearing potential not using adequate contraceptives or currently breastfeeding
* Life expectancy of less than twelve months
* Use of thrombectomy, artherectomy, cryoplasty, cutting balloon, drug-eluting balloon, embolic protection or laser devices during procedure
* Any patient considered to be hemodynamically unstable at onset of procedure
* Patient is currently participating in another investigational drug or device study that has not completed the entire follow up period.

Angiographic Exclusion Criteria

* Presence of an aortic thrombosis or significant common femoral ipsilateral stenosis
* Patients who exhibit persistent acute intraluminal thrombus of the proposed target lesion site
* Perforation, dissection or other injury of the access site or target vessel requiring additional stenting or surgical intervention prior to start of the index procedure
* Perforation at the angioplasty site evidenced by extravasation of contrast medium
* Aneurysm located at the level of the SFA and/or proximal popliteal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Major Adverse Event rate | 30 days post-procedure
  The primary safety endpoint of the study is the Major Adverse Event (MAE) rate at 30 days. MAE is defined as: clinically-driven target lesion revascularization, amputation of treated limb or all-cause mortality through 30 days post procedure.
Primary stent patency | 12 months post-procedure
  The primary effectiveness endpoint of the study is primary stent patency at 12 months. Primary patency is defined as absence of a hemodynamically significant stenosis on duplex ultrasound (systolic velocity ratio no greater than 2.4) at the target lesion and without TLR within 12 months.

SECONDARY OUTCOMES:
Technical success | 1 day post-procedure
  Technical success, defined as the ability to cross and stent the lesion, after predilation, and with or without additional post-dilation, and achieve residual angiographic stenosis no greater than 30%
Primary stent patency at 1 and 6 months | 1 and 6 months post-procedure
  Primary patency at 1, 6 months. Primary patency is defined as absence of a hemodynamically significant stenosis on duplex ultrasound (systolic velocity ratio no greater than 2.4) at the target lesion and without TLR within the time of procedure and the given follow-up.
Primary assisted patency | 1, 6 and 12 months post-procedure
  Primary assisted patency rate at 1, 6, 12-month follow-up. Defined as flow through the treated lesion maintained by repeat percutaneous intervention completed prior to complete vessel closure.
Secondary patency | 1, 6 and 12 months post-procedure
  Secondary patency rate at 1, 6, 12-month follow-up. Defined as flow through the treated lesion maintained by repeat percutaneous intervention after occlusion of the target lesion.
Target lesion revascularization | 12 months post-procedure
  Target lesion revascularization (TLR) is defined as a repeat intervention, within the study follow-up period of 12 months, to maintain or re-establish patency within the region of the treated arterial vessel plus 5 mm proximal and distal to the treated lesion edge.
limb-salvage | 12-months post-procedure
  Limb-salvage rate at all follow-up visits for the subgroup of patients with critical limb ischemia (Rutherford category 4), defined as absence of major amputation. Major amputation is defined as amputation at or above the ankle, as opposed to minor amputation, being an amputation at or below metatarsal level, preserving functionality of the foot)
Clinical success | 1, 6 and 12 months post-procedure
  Clinical success at follow-up, defined as an improvement of Rutherford classification at 1 day and 1, 6, 12-month follow-up of one class or more as compared to the pre-procedure Rutherford classification
Serious adverse events | 12-months post-procedure
  Serious adverse events defined as any clinical event that is fatal, life-threatening, or judged to be severe by the investigator; resulted in persistent or significant disability; necessitated surgical or percutaneous intervention; or required prolonged hospitalization.

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - Imelda Hospital, Bonheiden, Antwerp
  - University Hospital Antwerp, Edegem, Antwerp
  - A.Z. Sint-Blasius, Dendermonde, East-Flanders